CLINICAL TRIAL: NCT06257706
Title: An Interventional Study to Evaluate Treating to a Target of Transmural Healing in Patients With Moderately to Severely Active Crohn's Disease
Brief Title: VECTORS - A Study to Evaluate Transmural Healing as a Treatment Target in Crohn's Disease
Acronym: VECTORS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Alimentiv Inc. (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAK01769
Record Dates: First submitted 2024-01-24; First posted 2024-02-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Moderately to Severely Active Crohn's Disease; Crohn Disease; Disease Crohn
MeSH Terms: conditions — Crohn Disease | interventions — vedolizumab

STUDY DESIGN:
Intervention Model Description: This is an interventional, randomized, parallel-group, multicenter, controlled study. A total of approximately 304 participants with moderately-to-severely active CD from multiple international sites will be enrolled into this study. All qualified participants will be randomly assigned in a 1:1 ratio to one of 2 different treatment target groups: Group 1 will be treated over 48 weeks to achieve a target of corticosteroid-free IUS-based outcomes + clinical remission + biomarker remission. Group 2 will be treated over 48 weeks to achieve a target of corticosteroid-free clinical remission + biomarker remission. Randomization will be stratified by the following 3 baseline factors each with 2 levels: prior exposure (within the last 5 years of the screening date) to an approved biologic/small molecule for CD (yes or no), disease location (ileal or colonic), and disease duration (≤ 2 years or >2 years, based on date of diagnosis).
Masking Description: Study participants and investigators will be unblinded to the treatment target group assignment.
  Central readers performing the assessment of IUS, endoscopy, and histology assessments will be blinded to treatment target randomization, participant, treatment received, and timepoint which will be used to determine treatment escalation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1: Corticosteroid-free IUS-based outcomes + clinical remission + biomarker remission (Other): Group 1 will be treated over 48 weeks to achieve a target of corticosteroid-free IUS-based outcomes + clinical remission + biomarker remission. At Week 22 and 30, the IUS-based component of the target will be IUS response and at Week 38, the final treatment target will be TMH.
  Interventions: Biological: Vedolizumab
- Group 2: Corticosteroid-free clinical remission + biomarker remission. (Other): Group 2 will be treated over 48 weeks to achieve a target of corticosteroid-free clinical remission + biomarker remission.
  Interventions: Biological: Vedolizumab

INTERVENTIONS:
Biological: Vedolizumab — All participants will begin a vedolizumab induction regimen of 300 mg IV at Weeks 0, 2, 6, and 10 followed by vedolizumab 300 mg IV every 8 weeks starting at Week 14. Treatment may be modified at Weeks 22, 30, and/or 38 based on the results of the target assessment at each of these time points.

SUMMARY:
Transmural healing (TMH) is recognized as a potentially important measure of Crohn's disease (CD) activity but not a formal target. Observational studies suggest that TMH may be associated with better long-term outcomes. The study will evaluate TMH using noninvasive intestinal ultrasound (IUS), a patient-friendly technique that can be performed routinely in clinical practice. The aim of the study is to determine if treating to a target of corticosteroid-free (CS-free) IUS outcomes + clinical symptoms + biomarkers is superior to a target of clinical symptoms + biomarkers alone in achieving CS-free endoscopic remission measured by the Simple Endoscopic Score for Crohn's Disease (SES-CD).

Qualified participants will be randomly assigned in a 1:1 ratio to one of 2 different target treatment groups.

Group 1: Participants will be treated over 48 weeks to achieve a target of corticosteroid-free IUS-based outcomes + clinical remission + biomarker remission. At Week 22 and 30, the IUS-based component of the target will be IUS response and at Week 38, the final treatment target will be TMH. Group 2: Participants will be treated over 48 weeks to achieve a target of corticosteroid-free clinical remission + biomarker remission.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 to 80 years, inclusive, at the time of consent;
2. Moderately to severely active CD at baseline defined by a CDAI score of 220 to 450 inclusive and SES-CD, excluding the presence of narrowing component, ≥6 (or ≥4 for participants with isolated ileal disease);
3. BWT on IUS of >4.0 mm in the terminal ileum or any colonic segment (excluding the rectum) as assessed by the mean of 2 longitudinal and 2 cross-sectional measurements of the same segment;
4. Biologic-naïve or have previous exposure (within the last 5 years of the screening date) to no more than 1 advanced therapeutic compound (approved biologic or small molecule drug) for the treatment of their CD. Note: only approximately 15% to 30% of the enrolled population will have had prior exposure to an advanced therapeutic;
5. Participants may continue stable dose (initiated at least 4 weeks prior to Screening) of 5-ASA for CD;
6. Persons of childbearing potential must have a negative serum pregnancy test prior to randomization and must use a highly effective method of contraception throughout the study. Females unable to bear children must have documentation of such in the source records;
7. Able to participate fully in all aspects of this clinical trial;
8. Written informed consent must be obtained and documented.

Exclusion Criteria:

1. Current or previous treatment with vedolizumab, etrolizumab, or natalizumab;
2. Previously exposed to 2 or more compounds or classes of an advanced therapeutic compound (approved biologic or small molecule drug) for the treatment of their CD;
3. Change to oral corticosteroid therapy dosing within 2 weeks prior to randomization or a corticosteroid dose of >40 mg of prednisone or equivalent at randomization;
4. Only have inflammation proximal to the terminal ileum that cannot be reached by ileocolonoscopy;
5. Have a CD complication, such as symptomatic strictures in the small bowel with >3 cm prestenotic dilatation on any imaging modality, requiring procedural intervention;
6. Previous extensive colonic resection or missing >2 segments out of 5 (terminal ileum, right colon, transverse colon, sigmoid and left colon, and rectum), ileorectal anastomosis, or a proctocolectomy;
7. Ostomy or ileoanal pouch;
8. Short bowel syndrome;
9. Fibrotic-only stricture in the ileum or colon without evidence of active inflammation (in the investigator's judgment), including any impassable stenosis;
10. Abscess >2 cm, detected by IUS or endoscopy; participants with draining fistulas are not excluded;
11. Serious underlying disease other than CD that, in the opinion of the investigator, may interfere with the participant's ability to participate fully in the study or would compromise participant safety;
12. Positive stool test for Clostridioides difficile infection (as demonstrated by positive toxin);
13. Known HIV or hepatitis B or C infection. If a negative test result is available in the 12 months prior to randomization, retesting is not required;
14. Known active or latent tuberculosis (TB); if a negative test result is available in the 12 months prior to randomization, confirmatory testing (per standard of care) is not required before randomization;
15. Other systemic or opportunistic infection (including cytomegalovirus), any other clinically significant extraintestinal infection, or recurring infection within 6 months of randomization;
16. Has active cerebral/meningeal disease, signs, symptoms, or any history of progressive multifocal leukoencephalopathy (PML) prior to randomization;
17. Hypersensitivity, allergy, or intolerance to any excipient of vedolizumab or any other contraindication to vedolizumab;
18. Active severe infection such as sepsis, cytomegalovirus, listeriosis, or opportunistic infection.
19. Unwillingness to withhold protocol-prohibited medications during the trial;
20. Concurrent or previous participation in another clinical trial and received any investigational therapy within 30 days prior to randomization;
21. History of alcohol or drug abuse that in the opinion of the investigator may interfere with the participant's ability to comply with the study procedures;
22. Prior enrolment in the current study and had received study treatment;
23. Pregnant, lactating, or intending to become pregnant/impregnate a partner before, during, or within 18 weeks after the last dose; or intending to donate ova or sperm during such time period;
24. Vaccination with a live or live-attenuated vaccine within 4 weeks prior to randomization, or planned vaccination with a live or live-attenuated vaccine during participation in the study;
25. Any person performing mandatory military service, deprived of liberty, in a residential care setting, or any person who, due to a judicial decision, cannot take part in clinical studies;
26. The person is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (e.g., spouse, parent, child, sibling).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2029-01-03 (Estimated); Study Completion 2029-02-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with Corticosteroid-free Endoscopic remission in group 1 and group 2 at week 48 | week 48
  Corticosteroid-free is defined as not using corticosteroids at the time of the assessment. Endoscopic remission is defined by a total Simple Endoscopic Score for CD (SES-CD) ≤4 and at least a 2-point reduction versus baseline with no subscore greater than 1 in any individual variable. The SES-CD scores 4 endoscopic items (ulcer size, proportion of ulcerated surface, proportion of the surface area affected by any disease lesion, and stenosis) from 0 to 3, with higher scores representing more severe endoscopic disease activity. Each variable is scored for the 5 intestinal segments (ileum, right colon, transverse colon, left colon, and rectum) and summed to provide the total variable score. The sum of each variable score ranges from 0 to 15, except for stenosis (ranges from 0 to 11), because 3 represents a stenosis through which a colonoscope cannot be passed and therefore, can only be observed once. Total SES-CD score is then calculated by summing the item scores (range, 0-56 points).

SECONDARY OUTCOMES:
Percentage of participants with Corticosteroid-free Transmural healing (TMH)+Endoscopic remission+Clinical remission in group 1 and group 2 at week 48 | week 48
  Transmural healing is defined by Bowel wall thickness (BWT) ≤3.0 mm and color Doppler signal (CDS) 0 in all evaluable segments assessed by Intestinal Ultrasound.
  Endoscopic remission is defined by achievement of a total Simple Endoscopic Score for CD (SES-CD) ≤4 and at least a 2-point reduction versus baseline with no subscore greater than 1 in any individual variable. The SES-CD assesses 4 endoscopic variables: the size of ulcers, ulcerated surface, affected surface, and presence of narrowing. Each variable score ranging from 0 to 3. The total SES-CD score is calculated using the sum of all parameter scores in 5 segments: terminal ileum, right colon, transverse colon, left colon, and rectum.
  Clinical Remission is defined by achievement of Crohn's Disease Activity Index (CDAI) <150.
  CDAI consists of eight factors, each summed after adjustment with a weighting factor. Total score ranges from 0 to 600 points. Higher scores indicate more severity.
Percentage of participants with Corticosteroid-free IUS response+Endoscopic remission+Clinical Remission in group 1 and group 2 at week 48 | week 48
  IUS response is defined by reduction from baseline of 25% in Bowel Wall thickness (BWT) assessed by Intestinal Ultrasound (IUS).
  Endoscopic remission is defined by achievement of a total Simple Endoscopic Score for CD (SES-CD) ≤4 and at least a 2-point reduction versus baseline with no subscore greater than 1 in any individual variable.
  Clinical Remission is defined by achievement of Crohn's Disease Activity Index (CDAI) <150.
  The CDAI consists of 8 items including physical examination items, extraintestinal manifestations, the hematocrit, and PRO measures as recorded in the participant diary card for the 7 days prior to the clinic visit. Each item is multiplied by a weighting factor and summed to give a total CDAI score, ranging from 0 to over 600 points, with higher scores representing more severe disease activity.
Percentage of participants with Corticosteroid-free Endoscopic remission+Clinical Remission in group 1 and group 2 at week 48 | week 48
  Endoscopic remission is defined by achievement of a total Simple Endoscopic Score for CD (SES-CD) ≤4 and at least a 2-point reduction versus baseline with no subscore greater than 1 in any individual variable. The SES-CD scores 4 endoscopic items (ulcer size, proportion of ulcerated surface, proportion of the surface area affected by any disease lesion, and stenosis) from 0 to 3. Each variable is scored for the 5 intestinal segments (ileum, right colon, transverse colon, left colon, and rectum) and summed to provide the total variable score. Total SES-CD score is then summed up the item scores (range, 0-56 points).
  Clinical Remission is defined by Crohn's Disease Activity Index (CDAI) <150. CDAI consists of eight factors, each summed after adjustment with a weighting factor. Total score ranges from 0 to 600 points. Higher scores indicate more severity.
Percentage of participants with Corticosteroid-free endoscopic response+Clinical response in group 1 and group 2 at week 48 | week 48
  Endoscopic response is defined by Reduction in total Simple Endoscopic Score for CD (SES-CD) ≥50% from baseline. The SES-CD scores 4 endoscopic items (ulcer size, proportion of ulcerated surface, proportion of the surface area affected by any disease lesion, and stenosis) from 0 to 3, higher scores indicate more severity. Each variable is scored for the 5 intestinal segments (ileum, right colon, transverse colon, left colon, and rectum) and summed to provide the total variable score. The sum of each variable score ranges from 0 to 15, except for stenosis, where it ranges from 0 to 11. Total SES-CD score is then calculated by summing the item scores (range, 0-56 points).
  Clinical Response is defined by Crohn's Disease Activity Index (CDAI) decrease of ≥100 points from baseline. CDAI consists of eight factors, each summed after adjustment with a weighting factor. Total score ranges from 0 to 600 points. Higher scores indicate more severity.
Percentage of participants with Corticosteroid-free clinical remission in group 1 and group 2 at Week 14, Week 22 and Week 48. | week 14, week 22 and week 48
  Corticosteroid-free is defined as not using corticosteroids for treatment of CD at the time of the assessment.
  Clinical Remission is defined by achievement of Crohn's Disease Activity Index (CDAI) <150.
  The CDAI consists of 8 items including physical examination items, extraintestinal manifestations, the hematocrit, and PRO measures as recorded in the participant diary card for the 7 days prior to the clinic visit. Each item is multiplied by a weighting factor and summed to give a total CDAI score, ranging from 0 to over 600 points, with higher scores representing more severe disease activity.
Percentage of participants with Corticosteroid-free Clinical Response in group 1 and group 2 at week 14, week 22 and week 48 | week 14, week 22 and week 48
  Corticosteroid-free is defined as not using corticosteroids for treatment of CD at the time of the assessment.
  Clinical Response is defined by Crohn's Disease Activity Index (CDAI) decrease of ≥100 points from baseline. The CDAI consists of 8 items including physical examination items, extraintestinal manifestations, the hematocrit, and PRO measures as recorded in the participant diary card for the 7 days prior to the clinic visit. Each item is multiplied by a weighting factor and summed to give a total CDAI score, ranging from 0 to over 600 points, with higher scores representing more severe disease activity.
Crohn's Disease Activity Index(CDAI) total score and corresponding change from baseline during follow-up (Week 6, Week 14, Week 22, Week 30, Week 38, Week 48, Week 64, Week 80, Week 96) in group 1 and group 2 | week 6, week 14, week 22, week 30, week 38, week 48, week 64, week 80, week 96
  Crohn's Disease Activity Index (CDAI) consists of 8 items including physical examination items, extraintestinal manifestations, the hematocrit, and PRO measures as recorded in the participant diary card for the 7 days prior to the clinic visit. Each item is multiplied by a weighting factor and summed to give a total CDAI score, ranging from 0 to over 600 points, with higher scores representing more severe disease activity.
Percentage of participants with Corticosteroid-free endoscopic response in group 1 and group 2 at week 48 | week 48
  Corticosteroid-free is defined as not using corticosteroids for treatment of CD at the time of the assessment Endoscopic response is defined by Reduction in total Simple Endoscopic Score for CD (SES-CD) ≥50% from baseline. The SES-CD scores 4 endoscopic items (ulcer size, proportion of ulcerated surface, proportion of the surface area affected by any disease lesion, and stenosis) from 0 to 3, with higher scores representing more severe endoscopic disease activity. Each variable is scored for the 5 intestinal segments (ileum, right colon, transverse colon, left colon, and rectum) and summed to provide the total variable score. The sum of each variable score ranges from 0 to 15, except for stenosis, where it ranges from 0 to 11, because 3 represents a stenosis through which a colonoscope cannot be passed and therefore, can only be observed once. Total SES-CD score is then calculated by summing the item scores (range, 0-56 points).
SES-CD total score and corresponding change from baseline to Week 48 in group 1 and group 2 | week 48
  The SES-CD scores 4 endoscopic items (ulcer size, proportion of ulcerated surface, proportion of the surface area affected by any disease lesion, and stenosis) from 0 to 3, with higher scores representing more severe endoscopic disease activity. Each variable is scored for the 5 intestinal segments (ileum, right colon, transverse colon, left colon, and rectum) and summed to provide the total variable score. The sum of each variable score ranges from 0 to 15, except for stenosis, where it ranges from 0 to 11, because 3 represents a stenosis through which a colonoscope cannot be passed and therefore, can only be observed once. Total SES-CD score is then calculated by summing the item scores (range, 0-56 points).
Percentage of participants with Transmural healing (TMH) in group 1 and group 2 at week 48 | week 48
  Transmural Healing (TMH) is defined by Bowel wall thickness (BWT) ≤3.0 mm and color Doppler signal (CDS) 0 in all evaluable segments assessed by Intestinal Ultrasound
Percentage of participants with Intestinal Ultrasound (IUS) response in group 1 and group 2 at Week 48 | week 48
  IUS response is defined by reduction from baseline of 25% in Bowel Wall thickness (BWT) assessed by Intestinal Ultrasound (IUS)
Bowel Wall Thickness (BWT) measured by Intestinal Ultrasound (IUS) in mm and corresponding change from baseline at Week 48 in group 1 and group 2. | week 48
Color Doppler signal (CDS) and corresponding change from baseline at Week 48 in group 1 and group 2. | week 48
International Bowel Ultrasound Segmental Activity Score (IBUS-SAS) (per segment as well as total) and corresponding change from baseline at Week 48 in group 1 and group 2 | week 48
  International Bowel Ultrasound Segmental Activity Score (IBUS-SAS) is a 0-100 numerical activity index for Crohn's disease calculated from four Intestinal Ultrasound (IUS) parameters
Percentage of participants with Transmural healing (TMH) at week 14, week 22, week 30, week 38, and week 48 in group 1 | week 14, week 22, week 30, week 38, week 48
  Transmural Healing (TMH) is defined by Bowel wall thickness (BWT) ≤3.0 mm and color Doppler signal (CDS) 0 in all evaluable segments assessed by Intestinal Ultrasound
Percentage of participants with Intestinal Ultrasound (IUS) response at week 14, week 22, week 30, week 38, and week 48 in group 1 | week 14, week 22, week 30, week 38, week 48
  IUS response is defined by reduction from baseline of 25% in Bowel Wall thickness (BWT) assessed by Intestinal Ultrasound (IUS)
Bowel Wall Thickness (BWT) measured by Intestinal Ultrasound (IUS) in mm and corresponding change from baseline at week 14, week 22, week 30, week 38, and week 48 in group 1 | week 14, week 22, week 30, week 38, week 48
Color Doppler signal (CDS) and corresponding change from baseline at week 14, week 22, week 30, week 38, and week 48 in group 1 | week 14, week 22, week 30, week 38, week 48
International Bowel Ultrasound Segmental Activity Score (IBUS-SAS) (per segment as well as total) and corresponding change from baseline at week 14, week 22, week 30, week 38, and week 48 in group 1 | week 14, week 22, week 30, week 38, week 48
  International Bowel Ultrasound Segmental Activity Score (IBUS-SAS) is a 0-100 numerical activity index for Crohn's disease calculated from four Intestinal Ultrasound (IUS) parameters
Percentage of participants with Histologic remission at week 48 in group 1 and group 2 | week 48
  Histologic remission is defined by Robarts Histopathology Index (RHI) score ≤3 (per segment) with subscores of 0 for lamina propria neutrophils and 0 for neutrophils in epithelium, as scored by central reader.
  The RHI is a validated instrument that measures histologic disease activity and consists of 4 subscores (chronic inflammatory infiltrate, lamina propria neutrophils, neutrophils in epithelium, and erosion or ulceration). Each subscore ranges from 0-3, with higher subscores indicating greater histologic disease activity. The RHI score is calculated as: (1 x chronic inflammatory infiltrate) + (2 x lamina propria neutrophils) + (3 x neutrophils in epithelium) + (5 x erosion or ulceration). The RHI therefore ranges from 0-33, with higher scores indicating greater histologic disease activity.
Percentage of participants with Histologic response at week 48 in group 1 and group 2 | week 48
  Histologic response is defined as ≥7-point reduction from baseline in RHI, as scored by a central reader.
  The RHI is a validated instrument that measures histologic disease activity and consists of 4 subscores (chronic inflammatory infiltrate, lamina propria neutrophils, neutrophils in epithelium, and erosion or ulceration). Each subscore ranges from 0-3, with higher subscores indicating greater histologic disease activity. The RHI score is calculated as: (1 x chronic inflammatory infiltrate) + (2 x lamina propria neutrophils) + (3 x neutrophils in epithelium) + (5 x erosion or ulceration). The RHI therefore ranges from 0-33, with higher scores indicating greater histologic disease activity.
Percentage of patients with Biomarker remission at week 48, week 64, week 80 and week 96 in group 1 and group 2 | week 48, week 64, week 80, week 96
  Biomarker remission is defined as Normalization of C-reactive protein (CRP) <5 mg/mL and fecal calprotectin (FCal) <250 μg/g
Percentage of patients with Biomarker response at week 48, week 64, week 80 and week 96 in group 1 and group 2 | week 48, week 64, week 80, week 96
  Biomarker response is defined as ≥50% reduction from baseline in either C-reactive protein (CRP) or fecal calprotectin (FCal)
Percentage of participants with C-reactive protein (CRP) response during follow-up (Week 6, week 14, week 22, week 30, week 38, week 48, week 64, week 80 and week 96) in group 1 and group 2 | week 6, week 14, week 22, week 30, week 38, week 48, week 64, week 80, week 96
  C-reactive protein (CRP) response is defined by ≥50% reduction from baseline
Percentage of participants with fecal calprotectin (FCal) response during follow-up (Week 6, week 14, week 22, week 30, week 38, week 48, week 64, week 80 and week 96) in group 1 and group 2 | week 6, week 14, week 22, week 30, week 38, week 48, week 64, week 80, week 96
  Fecal calprotectin (FCal) response is defined by ≥50% reduction from baseline
Changes in C-reactive protein (CRP) from baseline during follow-up (Week 6, week 14, week 22, week 30, week 38, week 48, week 64, week 80 and week 96) in group 1 and group 2 | week 6, week 14, week 22, week 30, week 38, week 48, week 64, week 80, week 96
Changes in fecal calprotectin (FCal) from baseline during follow-up (Week 6, week 14, week 22, week 30, week 38, week 48, week 64, week 80 and week 96) in group 1 and group 2 | week 6, week 14, week 22, week 30, week 38, week 48, week 64, week 80, week 96
2-item Patient-Reported Outcome (PRO-2) score and corresponding changes from baseline during follow-up (Weeks 6, week 14, week 22, week 30, week 38, week 48, week 64, week 80 and week 96) in group 1 and group 2 | week 6, week 14, week 22, week 30, week 38, week 48, week 64, week 80, week 96
  The PRO-2 consists of the 2 CDAI component items: daily stool frequency and abdominal pain. Study participants record the number of liquid or very soft stools and rate abdominal pain (range, 0-3) daily in their participant diary for the 7 days prior to a clinic visit, excluding days of bowel preparation and ileocolonoscopy. The stool frequency and abdominal pain scores are calculated as the average scores over the 7-day period.
Symptoms and Impacts Questionnaire for CD (SIQ-CD) score and corresponding changes from baseline during follow-up (Weeks 6, week 14, week 22, week 30, week 38, week 48, week 64, week 80 and week 96) in group 1 and group 2 | week 6, week 14, week 22, week 30, week 38, week 48, week 64, week 80, week 96
  SIQ-CD tool consists of a symptom domain, which includes Gastrointestinal (GI), pain and discomfort, nutrition-related, and fatigue-related symptoms; and an impact domain, which includes concepts related to daily activities, nutrition, emotional well-being, and productivity.
Urgency Numerical Rating Score (NRS) and corresponding changes from baseline during follow-up (Weeks 6, week 14, week 22, week 30, week 38, week 48, week 64, week 80 and week 96) in group 1 and group 2 | week 6, week 14, week 22, week 30, week 38, week 48, week 64, week 80, week 96
  The Urgency NRS evaluates the participant's sense of urgency to have a bowel movement over the previous 24 hours and is rated on an 11-point Likert scale, from 0 for "no urgency" to 10 for "worst possible urgency"
Inflammatory Bowel Disease Questionnaire (IBDQ) score and corresponding changes from baseline during follow-up (Weeks 30, week 48 and week 96) in group 1 and group 2 | week 30, week 48, week 96
  The IBDQ measures health related quality of life in subjects with inflammatory bowel disease. It consists of 32 questions each with a graded response of 1 (worst) to 7 (best). The score ranges from 32 to 224
Time to CD-related complication from randomization through Week 96 in group 1 and group 2 | from randomization through Week 96
  CD-related complication will be defined as any of the following: (1) CD-related surgery; (2) CD-related hospitalization; (3) CD medication-related complication; (4) CD procedure-related complication; (5) Rescue therapy for a documented CD-related flare e.g., new initiation of an advanced therapy other than VDZ (approved biologic or small molecule), dose escalation of vedolizumab, or dose intensification beyond the dose used at randomization of a corticosteroid after Week 48 or; (6) Other CD-related complication
Time to each component of CD-related complication in group 1 and group 2 | from randomization through Week 96
Percentage of participants who switched to an alternate biologic (yes/no) by Week 48 and Week 96 | week 48, week 96
Exposure-adjusted incidence rates of serious adverse events (SAEs), all adverse events (AEs), and AEs of special interest (AESIs) in group 1 and group 2 | up to week 96
  Defined as the number of participants experiencing the event per 100 person-years (PYs) of exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Vipul Jairath, MD, Principal Investigator — Alimentiv Inc.
Locations (69):
- United States (3):
  - TLC Clinical Research Inc - Los Angeles, Los Angeles, California
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Houston Methodist Hospital, Houston, Texas
- Australia (10):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Mater Misericordiae Ltd, South Brisbane, Queensland
  - Calvary Adelaide Hospital, Adelaide, South Australia
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - Northern Hospital Epping, Epping, Victoria
  - Austin Health, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Harry Perkins institute of Medical Research - Fiona Stanley Hospital, Murdoch, Western Australia
- Belgium (6):
  - VITAZ - AZ Nikolaas, Sint-Niklaas, Antwerpen
  - Imelda Ziekenhuis Bonheiden, Bonheiden, Antwerp
  - University Hospital Ghent, Ghent, East Flanders
  - UZ Leuven-University Hospital Gasthuisberg, Leuven, Flemish Brabant
  - AZ Delta - Rumbeke Campus, Roeselare, West Flanders
  - ULB Hopital Erasme, Brussels
- Canada (6):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Dept of Medicine, Division of Gastroenterology, Edmonton, Alberta
  - Viable Clinical Research - Bridgewater, Bridgewater, Nova Scotia
  - LHSC - University Campus, London, Ontario
  - LHSC - Victoria Hospital, London, Ontario
  - Toronto Immune and Digestive Health Institute Inc. (TIDHI), Toronto, Ontario
- Czechia (2):
  - Vojenska nemocnice Brno, Brno, South Moravian
  - Fakultni Nemocnice Brno, Brno, South Moravian
- Denmark (8):
  - Herlev Hospital, Herlev, Capital Region
  - Nordsjaellands Hospital - Hillerod, Hillerød, Capital Region
  - Bispebjerg Hospital, Copenhagen NV, Capital
  - Hvidovre Hospital, Hvidovre, Capital
  - Aarhus Universitetshospital, Aarhus, Central Denmark
  - Randers Regional Hospital, Randers, Central Denmark
  - Sjaellands Universitets hospitall Koge, Køge, Region Sjælland
  - Svendborg Hospital, Svendborg
- France (3):
  - Hopital Lyon Sud, Pierre-Bénite, Auvergne-Rhône-Alpes
  - APHM, Marseille, Provence-Alpes-Côte d'Azur Region
  - Groupe Hospitalier Prive Ambroise Pare - Hartmann, Neuilly-sur-Seine
- Germany (5):
  - Universitatsklinikum Augsburg, Augsburg, Bavaria
  - Universitatsklinkum Frankfurt - Goethe Universitat, Frankfurt am Main, Hesse
  - Klinikum Luneburg, Lüneburg, Lower Saxony
  - Universitaetsklinikum Schleswig-Holstein (UKSH)- Campus Kiel, Kiel, Schleswig-Holstein
  - Universitats Klinikum Freiburg, Freiburg im Breisgau
- Italy (4):
  - Ospedale Casa Sollievo della Sofferenza IRCCS, San Giovanni Rotondo, Foggia
  - Ospedale Luigi Sacco, Milan, Lombardy
  - Ospedale San Raffaele S.r.I., Milan, Milan
  - Policlinico Universitario Agostino Gemelli, Roma, Rome
- Netherlands (4):
  - Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland
  - Amsterdam UMC - VU Medisch Centrum, Amsterdam, North Holland
  - Erasmus Medisch Centrum (MC), Rotterdam, South Holland
  - ETZ - St. Elisabeth Hospital, Tilburg
- Poland (11):
  - Oddzial Gastroenterologiczny SP ZOZ w Lecznej, Łęczna, Gmina Leczna
  - SOLUMED Centrum Medyczne, Poznan, Greater Poland Voivodeship
  - GASTROMED - Kopon, Zmudzinski I Wspolnicy Sp.j., Torun, Kuyavian-Pomeranian Voivodeship
  - Melita Medical Sp Zoo, Wroclaw, Lower Silesian Voivodeship
  - Bodyclinic Sp.z.o.o. Sp.K, Warsaw, Masovia
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw, Masovia
  - Centrum Medyczne Medyk, Rzeszów, Podkarpackie Voivodeship
  - Vita Longa Sp. z o.o., Katowice, Silesian
  - Sonomed Sp. z o.o. - Centrum Medyczne, Szczecin, West Pomerianian
  - Twoja Przychodnia-Centrum Medyczne Opole, Opole
  - EuroMediCare (EMC) Instytut Medyczny SA, Wroclaw
- LisbonCentro Hospitalar Lisboa Norte, EPE- Hospital de Santa Maria, Lisbon, Portugal
- United Kingdom (6):
  - Nottingham University Hospitals NHS Trust - QMC, Nottingham, East Midlands
  - London North West University Healthcare NHS Trust - Northwick Park Hospital, Harrow, Middlesex
  - Western General Hospital, Edinburgh
  - Barts Health NHS Trust - The Royal London Hospital, London
  - University College London Hospitals NHS Foundation Trust, London
  - Kings College Hospital NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the results reported in this article may be made available upon reasonable request, subject to review and approval by the study sponsor, execution of a data use agreement, and in accordance with participant consent and applicable privacy and data protection requirements.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: 06JAN2026 - 31JAN2029
Access Criteria: De-identified individual participant data underlying the results reported in this article may be made available upon reasonable request, subject to review and approval by the study sponsor, execution of a data use agreement, and in accordance with participant consent and applicable privacy and data protection requirements.